CLINICAL TRIAL: NCT05097378
Title: Perioperative Encorafinib+Binimetinib in BRAFV600 Mutant Clinically Detected AJCC Stage III (B/C/D) or Oligometastatic Stage IV Melanoma
Brief Title: Perioperative Encobini in BRAFV600 Mutant Stage III (B/C/D) or Oligometastatic Stage IV Melanoma
Acronym: PREMIUM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREMIUM
Record Dates: First submitted 2021-10-04; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Melanoma; Cancer
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — encorafenib; binimetinib

STUDY DESIGN:
Intervention Model Description: Neoadjuvant and adjuvant administration schedule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EncoBini Arm (Experimental): Oral encorafenib 450mg once daily and oral binimetinib 45mg twice daily for 8 weeks pre-operative and for up to 44 weeks post-operative.
  Interventions: Drug: Encorafenib + Binimetinib
- Standard Arm (Active Comparator): Immediate surgery followed by Investigator's choice of standard adjuvant therapy to commence within 12 weeks of surgery and to continue for up to 52 weeks.
  Interventions: Drug: Standard Adjuvant Treatment

INTERVENTIONS:
Drug: Encorafenib + Binimetinib — Encorafenib is a potent and highly selective ATP-competitive small molecule RAF kinase inhibitor, which suppresses the RAF/MEK/ERK pathway in tumour cells expressing several mutated forms of BRAF kinase (V600E, D and K).
  Binimetinib is an ATP-uncompetitive, reversible inhibitor of the kinase activity of mitogen-activated extracellular signal regulated kinase 1 (MEK1) and MEK2. Binimetinib inhibits activation of MEK by BRAF and inhibits MEK kinase activity
  Other Names: Braftovi + Mektovi
  Arms: EncoBini Arm
Drug: Standard Adjuvant Treatment — Standard Adjuvant Treatment
  Arms: Standard Arm

SUMMARY:
A two-arm, randomised trial investigating the response of encorafenib and binimetinib compared to standard adjuvant therapy.

DETAILED DESCRIPTION:
A phase II, multi-centre, open label, randomised trial.

The trial will assess the delivery, response rate, treatment compliance, efficacy and safety of encorafenib and binimetinib compared to standard adjuvant therapy in patients with BRAFV600 mutant clinically detected AJCC stage III(B/C/D) or oligometastatic stage IV Melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate
* Aged ≥ 18 years old
* AJCC 8th edition stage III (B/C/D), or extracranial oligometastatic stage IV BRAFV600 mutant melanoma, based on histological/cytological and radiological assessments for which surgery is planned, and resection is expected to remove all known tumour(s) with R0 resection margins. 'Oligometastatic stage IV' is defined for the purpose of this trial as M stage disease confined to a single body organ excluding the brain that can be readily removed surgically with anticipated clear margins
* For stage III patients, confirmation of no evidence of distant metastatic disease using preferred imaging modalities including CT body or PET/CT and CT or MRI head
* For stage IV patients, confirmation of no evidence of unresectable metastatic disease, or metastatic disease in more than 1 body organ, using preferred imaging modalities including CT body or PET/CT and CT or MRI head. The site of metastasis should not be in bone, or CNS, or in any other body site where complete resection is not feasible
* The planned resectable disease must be radiologically measurable using standard imaging modalities.
* Baseline tumour assessments must be done within 28 days prior to randomisation
* BRAF V600E or V600K mutation confirmation
* Received no prior BRAF or MEK inhibitors
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Predicted life expectancy >12 months
* Normal QTc interval (<480msec) on ECG and left ventricular ejection fraction within normal limits, assessed by echocardiogram or MUGA
* Adequate bone marrow function defined as:
* Absolute neutrophil count (ANC) ≥1.5 x 109 /L
* Haemoglobin (Hb) ≥ 90 g/L
* Platelets ≥100 x 109 /L
* Adequate liver function defined as:
* Aspartate aminotransferase (AST) and/or alanine transaminase (ALT) ≤2.5 x upper limit of normal range (ULN)
* Total bilirubin <1.5 x ULN (except if the patient has Gilbert Syndrome or liver metastases, in which case the bilirubin must be <3 x ULN)
* Adequate renal function defined as:
* a serum creatinine ≤1.5 x ULN or
* calculated creatinine clearance by Cockcroft-Gault of ≥40 mL/min
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, completion of QoL and PROM questionnaires and other procedures described in the protocol
* Women of child-bearing potential (WCBP) and all sexually active male patients must agree to use effective contraception methods throughout treatment
* Be able to swallow the trial medication
* Confirmation of adequate diagnostic tumour tissue available for research studies

Exclusion criteria

* Prior adjuvant therapy for resected primary or loco-regional melanoma
* Other invasive malignancies diagnosed within the last 2 years which are not in complete remission, or for which additional therapy is required
* Brain or bone metastases
* Non-cutaneous primary site of melanoma
* Prior radiotherapy to the site planned for surgery
* History or current evidence of retinal vein occlusion (RVO) or risk factors for RVO (uncontrolled glaucoma, ocular hypertension, history of hyperviscosity, or hypercoagulability syndromes)
* Left ventricular function <50%
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the investigator would place the patient at undue risk or interfere with the trial. Examples include, but are not limited to:
* Patients with uncontrolled ischaemic heart or other cardiovascular event (myocardial infarction (MI), new angina, stroke transient ischaemic attack (TIA), or new congestive cardiac failure (CCF)) within the last 6 months
* Uncontrolled hypertension
* Patients with stable but significant cardiovascular disease defined by heart failure (New York Heart Association Functional Classification (NYHF) III or IV or frequent angina
* Patients with baseline QTC interval > 480 msec on electrocardiogram (ECG)
* Left ventricular ejection fraction below the lower limit of normal
* Presence of active infection
* Cirrhotic liver disease, known chronic active or acute hepatitis B, or hepatitis C
* Known allergy or hypersensitivity to Encorafenib or Binimetinib, or their excipients. Binimetinib contains lactose, so patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption will be excluded.
* Women who are pregnant, plan to become pregnant or are lactating during the trial period
* Use of any other investigational anti-cancer drugs (a washout period of 28 days would be required)
* Use of strong inducers and inhibitors of CYP3A4 (Appendix 4 - Prohibited Medication)
* Known HIV or active Hep B or Hep C infection
* Patients who have neuromuscular disorders associated with elevated creatine phosphokinase (CK, e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Autoimmune conditions requiring regular or intermittent use of any systemic steroid or immunosuppressive drugs, with the exception of steroid inhalers
* Any immunotherapy in the last 3 months
* Prior radiotherapy to the site of disease planned for resection
* Concurrent participation in an interventional clinical trial (observational studies allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | During scheduled surgery
  % of patients with a complete response using Haemotoxylin and Eosin staining of tumour removed at surgery.

SECONDARY OUTCOMES:
Treatment compliance | Through study completion for an average of 12 months
  Incidence of missed treatment doses assessed from number of tablets returned.
Radiological response | Through study completion for an average of 12 months
  % of patients with a complete response using CT scan tumour measurement assessment (RECIST) from start of treatment until 8 weeks.
Toxicity of treatment | Through study completion for an average of 12 months
  Rate of patients with drug related toxicities reported from start of study until end of treatment
Lymphoedema toxicity | Through study completion for an average of 12 months
  Incidence of lymphoedema toxicity using circumferential limb measurement and questionnaires for an average of 12 months.
Survival rate | Through study completion for an average of 12 months
  Number of patients deceased from start of treatment for an average of 12 months.
Quality of life | Through study completion for an average of 12 months
  Quality of life assessed by Functional Assessment of Cancer Therapy - Melanoma (FACT-M) questionnaire for an average of 12 months.
Recruitment rate | Through study completion for an average of 12 months
  Rate of monthly recruitment achieved during the last 6 months of the trial recruitment period

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No